CLINICAL TRIAL: NCT07185971
Title: PAVE (Parallactic Visual-Field Enhancement) System for Treatment of Chronic Visual Field Loss
Brief Title: PAVE (Parallactic Visual-Field Enhancement) System for Treatment of Chronic Visual Field Loss Due to Stroke, Traumatic Brain Injury, or Brain Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroAEye LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN001
Record Dates: First submitted 2025-09-11; First posted 2025-09-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Homonymous Hemianopsia; Homonymous Quadrantanopia
Keywords: PAVE; Parallactic Visual-Field Enhancement; NeuroAEye; chronic visual field loss
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Intervention Model Description: Random Controlled Trial with blinding of investigators and subjects.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Test (Experimental): Weekly treatment using actual PAVE therapy software operating on a virtual reality head mounted display.
  Interventions: Device: PAVE (Parallactic Visual-Field Enhancement) treatment using a virtual reality head mounted display
- Control (Placebo Comparator): Weekly treatment using a placebo that include PAVE software absent the functional component, operating on a virtual reality head mounted display.
  Interventions: Device: PAVE Placebo

INTERVENTIONS:
Device: PAVE (Parallactic Visual-Field Enhancement) treatment using a virtual reality head mounted display — PAVE (Parallactic Visual-Field Enhancement) treatment is visual stimulation using a virtual reality head mounted display. The treatment is weekly and entails two 7 minute session separated by a minimum 1 minute intermission. The actual therapy is preceded by a visual field assessment and is followed by a second visual field assessment.
  Arms: Test
Device: PAVE Placebo — The placebo uses the same PAVE software but the functional aspect of the software that is intended to produce the effect in the test group is absent.
  Arms: Control

SUMMARY:
This is a research study to evaluate the effectiveness of the PAVE (Parallactic Visual-Field Enhancement) System for the treatment of chronic visual field loss due to stroke, traumatic brain injury, or brain surgery. The PAVE regimen involves the use of a virtual reality headset to deliver visual stimulation to subjects diagnosed with visual field loss.

The primary objective is to demonstrate that the clinical outcomes from exposure to the PAVE therapy (test group) are statistically superior to those achieved with a placebo (control group). The primary outcome is an increase in visual field area as measured with Goldmann-type kinetic perimetry.

The secondary outcome will be demonstration that the subjective assessment of visual function using the National Eye Institute Visual Function Questionnaire (NEI-VFQ) is better for the test group when compared with the control group.

The participants will visit the investigators office once per week for a minimum of eight weeks and a maximum of twenty four weeks and receive a therapy session. Every four weeks the participants visual field will be measured using kinetic perimetry. Every eight weeks the participant will complete the NEI-VFQ. Four weeks after the completion of the therapy sessions a follow up visit will take place where visual field measurement using kinetic perimetry and NEI-VFQ will be administered.

DETAILED DESCRIPTION:
This clinical investigation will focus on patients with chronic visual field loss following a cerebrovascular accident (CVA), a traumatic brain injury (TBI), or surgery of the brain. The CVA and TBI and some surgeries of the brain may affect bilateral visual fields (homonymous hemianopia, quadrantanopia, or general constriction). While perimetric visual field improvements can occur spontaneously in the first few months after brain injury, after six months the condition is considered chronic and permanent .

This study will include patients at least 6 months after the brain injury event and up to five years after onset. If available for the study, patients suffering field loss as a result of brain surgery may also be enrolled. All patients shall have a definitive diagnosis of homonymous hemianopia, quadrantanopia, or general constriction. The patients shall have the ability to wear the HMD for a 30-minute session performed in the clinic at least once per week. Patients will be between 21 and 80 years of age. The clinical study shall be a random controlled trial with the test group receiving therapy with the PAVE software on the HMD. The control group will receive placebo treatment using the HMD. The placebo software will replace the patterns of PAVE with a different pattern. In both the control and test groups the patient is requested to focus on the central target during the session. The initial sample size will be n=15 for each group. Performance will be evaluated using a semiautomated kinetic perimeter (SKP) measurement derived from the Goldmann method. The study will be an adaptive design with interim data analysis and hypotheses evaluation performed every four weeks after the subjects have completed that week's therapy. Termination of therapy may occur four weeks after the interim data assessment. The decision to end the study will depend on the variance and the rate of change in the perimetry measures. If the rate of improvement of the test group appears constant, then the study will continue for at least another four weeks. If the variance between subjects is high, additional subjects may be recruited and added to the study to improve statistical power. The maximum duration of the study for an individual participant shall be 24 weeks of treatment and a 4 week follow-up for a total of 28 to 30 weeks.

The goal will be to demonstrate a statistically significant difference in the improvement of the visual field between the test and control groups. Additional endpoints will include the percentage of test group patients showing improvement compared with the mean of the control group and subjective assessment of the subject's visual performance using the National Eye Institute Visual Functioning Questionnaire (NEI-VFQ).

ELIGIBILITY:
Inclusion Criteria:

* This study will include patients at least 6 months after the CVA or TBI or brain surgery event and up to five (5) years after onset
* The patients shall have a definitive diagnosis of homonymous hemianopia or quadrantanopia or generalized constriction.

Exclusion Criteria:

* Presence of any physical, neurological, or mental disability that would interfere with receiving the therapy.
* Concurrent use of another visual therapy
* Concurrent use of medications judged to affect training (amphetamines, dopamine, etc.)
* Presence of ocular or neurological conditions that would interfere with training or cause a visual impairment including no residual vision, disorders of the eye, non-optic nerve heteronymous visual field defects
* Insufficient fixation ability
* Use of life supporting external medical device such as infusion pumps, ventricular assist devices, etc.
* Presence of active implantable medical device including but not limited to cardiac pacemakers, defibrillators, nerve stimulators, cochlear implants, etc.
* Subjects with known photosensitive epilepsy.
* Subjects with chronic active infections on the head and face should be excluded from the study
* Patients with known immune disorders for whom an infection could be life threatening should be excluded from the study.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Population Mean Change in Visual Field Area | Visual field area will be assessed at the baseline, week 4, week 8, week 12, week 16, week 20, week 24, and at the follow up at week 28.
  The visual field area is derived from the isopter plot output of semiautomated kinetic perimetry. A baseline visual field area will be taken and subsequent measurements will be compared to the baseline.

SECONDARY OUTCOMES:
Proportion of test group showing improvement. | The proportion of the test group showing improvement will be assessed at the conclusion of the study or week 28, whichever occurs first.
  The percentage of the test group that demonstrates improvement when compared to the mean change in field of view area for the control group.

OTHER OUTCOMES:
Change in Subjective Visual Function | NEI-VFQ will be administered at baseline, at week 8, week 16, week 24 and again at the 4 week post-treatment follow up which is week 28 if the study does not conclude earlier.
  Use of NEI-VFQ to survey subjects at baseline and intermediate endpoints with regard to their assessment of visual function. Compare baseline and final assessments.

CONTACTS AND LOCATIONS:
Overall Officials: DeAnn Fitzgerald, Doctor of Optometry, Principal Investigator — Dr. D. M. Fitzgerald & Associates
Locations (1):
- Dr. D. M. Fitzgerald & Associates, Cedar Rapids, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zahid S, Peeler C, Khan N, Davis J, Mahmood M, Heckenlively JR, Jayasundera T. Digital quantification of Goldmann visual fields (GVFs) as a means for genotype-phenotype comparisons and detection of progression in retinal degenerations. Adv Exp Med Biol. 2014;801:131-7. doi: 10.1007/978-1-4614-3209-8_17. PMID 24664690
- [Background] Pe'er J, Zajicek G, Barzel I. Computerised evaluation of visual fields. Br J Ophthalmol. 1983 Jan;67(1):50-3. doi: 10.1136/bjo.67.1.50. No abstract available. PMID 6848135
- [Background] Barry MP, Bittner AK, Yang L, Marcus R, Iftikhar MH, Dagnelie G. Variability and Errors of Manually Digitized Goldmann Visual Fields. Optom Vis Sci. 2016 Jul;93(7):720-30. doi: 10.1097/OPX.0000000000000869. PMID 27058594
- [Background] Christoforidis JB. Volume of visual field assessed with kinetic perimetry and its application to static perimetry. Clin Ophthalmol. 2011;5:535-41. doi: 10.2147/OPTH.S18815. Epub 2011 Apr 26. PMID 21573042
- [Background] Bittner AK, Iftikhar MH, Dagnelie G. Test-retest, within-visit variability of Goldmann visual fields in retinitis pigmentosa. Invest Ophthalmol Vis Sci. 2011 Oct 11;52(11):8042-6. doi: 10.1167/iovs.11-8321. PMID 21896857
- [Background] Rowe FJ, Hepworth LR, Hanna KL, Mistry M, Noonan CP. Accuracy of kinetic perimetry assessment with the Humphrey 850; an exploratory comparative study. Eye (Lond). 2019 Dec;33(12):1952-1960. doi: 10.1038/s41433-019-0520-1. Epub 2019 Jul 22. PMID 31332292
- [Background] Barnes CS, Schuchard RA, Birch DG, Dagnelie G, Wood L, Koenekoop RK, Bittner AK. Reliability of Semiautomated Kinetic Perimetry (SKP) and Goldmann Kinetic Perimetry in Children and Adults With Retinal Dystrophies. Transl Vis Sci Technol. 2019 Jun 11;8(3):36. doi: 10.1167/tvst.8.3.36. eCollection 2019 May. PMID 31211001
- [Background] Goodwin D. Homonymous hemianopia: challenges and solutions. Clin Ophthalmol. 2014 Sep 22;8:1919-27. doi: 10.2147/OPTH.S59452. eCollection 2014. PMID 25284978
- [Background] Grunda T, Marsalek P, Sykorova P. Homonymous hemianopia and related visual defects: Restoration of vision after a stroke. Acta Neurobiol Exp (Wars). 2013;73(2):237-49. doi: 10.55782/ane-2013-1933. PMID 23823985
- [Background] Bouwmeester L, Heutink J, Lucas C. The effect of visual training for patients with visual field defects due to brain damage: a systematic review. J Neurol Neurosurg Psychiatry. 2007 Jun;78(6):555-64. doi: 10.1136/jnnp.2006.103853. Epub 2006 Nov 29. PMID 17135455
- [Background] Gall C, Sabel BA. Reading performance after vision rehabilitation of subjects with homonymous visual field defects. PM R. 2012 Dec;4(12):928-35. doi: 10.1016/j.pmrj.2012.08.020. Epub 2012 Nov 2. PMID 23122896
- [Background] Poggel DA, Mueller I, Kasten E, Bunzenthal U, Sabel BA. Subjective and objective outcome measures of computer-based vision restoration training. NeuroRehabilitation. 2010;27(2):173-87. doi: 10.3233/NRE-2010-0594. PMID 20871147
- [Background] Kasten E, Bunzenthal U, Sabel BA. Visual field recovery after vision restoration therapy (VRT) is independent of eye movements: an eye tracker study. Behav Brain Res. 2006 Nov 25;175(1):18-26. doi: 10.1016/j.bbr.2006.07.024. Epub 2006 Sep 12. PMID 16970999
- [Background] Mueller I, Mast H, Sabel BA. Recovery of visual field defects: a large clinical observational study using vision restoration therapy. Restor Neurol Neurosci. 2007;25(5-6):563-72. PMID 18334773
- [Background] Gall C, Mueller I, Gudlin J, Lindig A, Schlueter D, Jobke S, Franke GH, Sabel BA. Vision- and health-related quality of life before and after vision restoration training in cerebrally damaged patients. Restor Neurol Neurosci. 2008;26(4-5):341-53. PMID 18997310
- [Background] Poggel DA, Kasten E, Sabel BA. Attentional cueing improves vision restoration therapy in patients with visual field defects. Neurology. 2004 Dec 14;63(11):2069-76. doi: 10.1212/01.wnl.0000145773.26378.e5. PMID 15596752
- [Background] I. Mueller, D. Poggel, S. Kenkel, E. Kasten and B. A. Sabel, "Vision Restoration Therapy (VRT) after brain damage: subjective improvements of activities of daily life and their relationship to visual field enlargements.," Visual Impairment Research, vol. 5, no. 3, pp. 157-178, 2003.
- [Background] Marshall RS, Ferrera JJ, Barnes A, Xian Zhang, O'Brien KA, Chmayssani M, Hirsch J, Lazar RM. Brain activity associated with stimulation therapy of the visual borderzone in hemianopic stroke patients. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):136-44. doi: 10.1177/1545968307305522. Epub 2007 Aug 14. PMID 17698955
- [Background] Plow EB, Obretenova SN, Fregni F, Pascual-Leone A, Merabet LB. Comparison of visual field training for hemianopia with active versus sham transcranial direct cortical stimulation. Neurorehabil Neural Repair. 2012 Jul-Aug;26(6):616-26. doi: 10.1177/1545968311431963. Epub 2012 Jan 30. PMID 22291042
- [Background] Romano JG, Schulz P, Kenkel S, Todd DP. Visual field changes after a rehabilitation intervention: vision restoration therapy. J Neurol Sci. 2008 Oct 15;273(1-2):70-4. doi: 10.1016/j.jns.2008.06.026. Epub 2008 Jul 30. PMID 18672255
- [Background] Julkunen L, Tenovuo O, Jaaskelainen S, Hamalainen H. Rehabilitation of chronic post-stroke visual field defect with computer-assisted training: a clinical and neurophysiological study. Restor Neurol Neurosci. 2003;21(1-2):19-28. PMID 12808199
- [Background] Sabel BA, Kenkel S, Kasten E. Vision restoration therapy (VRT) efficacy as assessed by comparative perimetric analysis and subjective questionnaires. Restor Neurol Neurosci. 2004;22(6):399-420. PMID 15798360
- [Background] Kasten E, Wust S, Behrens-Baumann W, Sabel BA. Computer-based training for the treatment of partial blindness. Nat Med. 1998 Sep;4(9):1083-7. doi: 10.1038/2079. PMID 9734406
- [Background] Kasten E, Sabel BA. Visual field enlargement after computer training in brain-damaged patients with homonymous deficits: an open pilot trial. Restor Neurol Neurosci. 1995 Jan 1;8(3):113-27. doi: 10.3233/RNN-1995-8302. PMID 21551894
- [Background] W. Padula, R. Munitz and W. M. Magrun, Neuro-Visual Processing Rehabilitation, Santa Ana, CA: Optometric Extension Program Foundation, 2012.
- [Background] R. Sanet and L. Press, "Spatial Vision," in Vision Rehabilitation: Multidisciplinary Care of the Patient Following Brain Injury, Boca Raton, FL, CRC Press, Taylor & Francis Group, 2011, pp. 77-152.
- [Background] Padula WV, Capo-Aponte JE, Padula WV, Singman EL, Jenness J. The consequence of spatial visual processing dysfunction caused by traumatic brain injury (TBI). Brain Inj. 2017;31(5):589-600. doi: 10.1080/02699052.2017.1291991. Epub 2017 Apr 25. PMID 28440687
- [Background] Saionz EL, Tadin D, Melnick MD, Huxlin KR. Functional preservation and enhanced capacity for visual restoration in subacute occipital stroke. Brain. 2020 Jun 1;143(6):1857-1872. doi: 10.1093/brain/awaa128. PMID 32428211